CLINICAL TRIAL: NCT04316988
Title: Ultrasonography Imaging Versus Waveform Capnography in Detecting Endotracheal Tube Placement During Intubation in a Tertiary Hospital.
Brief Title: Ultrasonography Versus Capnography in Detecting Endotracheal Tube Placement During Intubation in a Tertiary Hospital.
Status: Completed | Type: Observational
Sponsor: Tribhuvan University, Nepal (Other)
Responsible Party: Principal Investigator, Shirish Shakti Maskay, Dr, Tribhuvan University, Nepal
Other Study IDs: IOM
Record Dates: First submitted 2020-03-13; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Intubation; Ultrasound Imaging; Capnography
Keywords: Endotracheal intubation; Ultrasonography; Capnography
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ultrasonography: Ultrasonography group in whom after endotracheal intubation, the endotracheal tube position was confirmed by ultrasound machine over the trachea.
  Interventions: Diagnostic Test: Ultrasonography
- Capnography: Capnography group in whom after endotracheal intubation, the endotracheal tube position was confirmed by capnograph, evaluationg the graph character and end tidal CO2 value.

INTERVENTIONS:
Diagnostic Test: Ultrasonography — A real time 2D ultrasound evaluation was done over the trachea of the patient.
  Groups: Ultrasonography

SUMMARY:
After endotracheal intubation verifying the location of endotracheal tube is of utmost importance. Many methods have been applied but none is perfect. The standard practice in the investigator's center has been to use auscultation of chest with capnography.

Ultrasound machines are now gaining popularity and their access extends from operation theatres, emergency rooms and even many primary health centres. Both capnography and ultrasonography are safe.

This study found out that Ultrasonography and waveform capnography are both reliable methods of confirming endotracheal tube position. The use of ultrasound could help reduce time and increase precision of confirming endotracheal tube position. Ultrasound can confirm endotracheal tube position before manual bag ventilations, and thus may prevent aspiration of gastric contents into patient's lungs.

DETAILED DESCRIPTION:
This was a prospective, observational study conducted at the Tribhuvan University Teaching Hospital (TUTH) and Manmohan Cardiothoracic Vascular and Transplant Center (MCVTC) operating rooms from January 2017 to July 2017. Ethical approval from the Institutional Review Board (IRB) of Institute of Medicine (IOM) and the Department of Anaesthesiology, Maharajgunj Medical College (MMC) was taken. Written informed consent was taken.

ASA I and II patients over 16 years of age were included in this study. Patients with difficult airway and anticipated difficult intubation, respiratory diseases, poor functional status, emergency case, and patients at risk of aspiration were excluded.

The diagnostic characteristics of real-time, suprasternal, transtracheal ultrasonography and capnography were tested by calculating their respective sensitivities, specificities, positive predictive values (PPV), negative predictive values (NPV), accuracies and likelihood ratios. Comparison of time taken for confirmation of endotracheal tube position from the beginning of laryngoscopy, by ultrasonography versus capnography was done using t-statistics.

The degree of agreement of result between ultrasonography and capnography was tested with kappa statistics.

Out of the 95 patients studied, 11 had oesophageal intubation (Incidence of 11.57%). The overall accuracy of both ultrasonography and capnography was 96.84%. The sensitivity, specificity, PPV, NPV with their corresponding 95% confidence intervals (CI) for ultrasonography were 97.62% (91.66% - 99.71%), 90.91% (58.72% - 99.77%), 98.80% (92.67% - 99.81%), 83.33% (55.66% - 95.22%) respectively; and that for capnography were 96.43% (89.92% - 99.26%), 100% (71.51% - 100%), 100% (100% - 100%) and 78.57% (54.69% - 91.76%) respectively.

The likelihood ratio of a positive and a negative result for ultrasonography were 10.74 and 0.03 respectively, and that for capnography were infinity and 0.04 respectively.

The kappa value was 0.749 (95% CI: 0.567 - 0.931) which meant a good degree of agreement of result between these two methods.

The average time taken for confirmation of endotracheal tube by ultrasonography and capnography were 26.79 ± 7.64 seconds and 43.03 ± 8.71 seconds (mean ± standard deviation) respectively. The median time for confirmation was 26 seconds with interquartile range [15 - 37] seconds for ultrasonography and 42 seconds with interquartile range [29 - 55] seconds for capnography. Ultrasonography was found to be faster than capnography by 16.36 ± 3.23 seconds (mean ± standard deviation) and the difference in time was significant (p = 0.011).

During the study, one patient had unanticipated difficult intubation, and four had hypotension after induction of anaesthesia. These patients were excluded from the study and no sequalae of hypotension was seen in the patients, or no hypoxemia occured in the patient with unanticipated difficult intubation.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II patients of both sexes above 16 years of age undergoing general anaesthesia with endotracheal tube placement.

Exclusion Criteria:

* - Patient refusal
* ASA physical status III and above
* History of prior difficult bag and mask ventilation or difficult intubation
* History of prior oro-nasal or neck injuries, burns or scars
* Active oral, pharyngeal or tracheal infection or inflammatory changes
* Anticipated difficult airway or difficult intubation during preanaesthetic examination, with Mallampati grades II and above
* Lung parenchymal and pleural diseases. Examples: asthma, COPD, bronchiectasis, reactive lung diseases, pneumonia, tuberculosis, pleural effusion, pneumothorax, lung or pleural malignancy etc.
* Emergency surgery

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: American Society of Anesthesiologist classified status I and II patients from Nepalsese population, without any selection for gender, caste or ethnicity, and above 16 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
ULTRASONOGRAPHY IMAGING VERSUS WAVEFORM CAPNOGRAPHY IN DETECTING ENDOTRACHEAL TUBE PLACEMENT DURING INTUBATION IN A TERTIARY HOSPITAL | 6 months
  Ultrasonography and waveform capnography are both reliable and accurate methods of confirming endotracheal tube position

SECONDARY OUTCOMES:
Ultrasonography compared to capnography for confirming the endotacheal tube position after intuabtion | 6 months
  * Using real-time transtracheal ultrasound can help confirm endotracheal tube position earlier than capnography.
  * Using real-time transtracheal ultrasound will help avoid manual bag ventilations to confirm endotracheal tube position and can prevent aspiration of gastric contents into lungs in cases of oesophageal intubation.

CONTACTS AND LOCATIONS:
Overall Officials: BISHWAS PRADHAN, MD, FCTA, Study Chair — Manmohan Cardiothoracic Vascular and Transplant Center, IOM; NINADINI SHRESTHA, MD, FIPM, Study Director — TU Teaching Hospital, IOM; PRISKA BASTOLA, MD, Study Director — Manmohan Cardiothoracic Vascular and Transplant Center, IOM

IPD SHARING:
Plan to Share IPD: Yes
Excel worksheet of patients data log entry includes age, sex and type of surgery; without disclosing personal patient details.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Indefinite
Access Criteria: email

REFERENCES:
- [Background] Rudraraju P, Eisen LA. Confirmation of endotracheal tube position: a narrative review. J Intensive Care Med. 2009 Sep-Oct;24(5):283-92. doi: 10.1177/0885066609340501. Epub 2009 Aug 3. PMID 19654121
- [Background] Wojtczak JA, Cattano D. Laryngo-tracheal ultrasonography to confirm correct endotracheal tube and laryngeal mask airway placement. J Ultrason. 2014 Dec;14(59):362-6. doi: 10.15557/JoU.2014.0037. Epub 2014 Dec 30. PMID 26672974
- [Background] Kundra P, Mishra SK, Ramesh A. Ultrasound of the airway. Indian J Anaesth. 2011 Sep;55(5):456-62. doi: 10.4103/0019-5049.89868. PMID 22174461
- [Background] Hajian-Tilaki K. Sample size estimation in diagnostic test studies of biomedical informatics. J Biomed Inform. 2014 Apr;48:193-204. doi: 10.1016/j.jbi.2014.02.013. Epub 2014 Feb 26. PMID 24582925
- [Background] Hagberg CA, Artime CA. Airway Management in the Adult. In: Miller RD, Cohen NH, Eriksson LI, Fleisher LA, Wiener-Kronish JP, Young WL, editors. Miller's Anesthesia. 8th ed. Philadelphia: Elsevier Saunders; 2015. p. 1665-6.
- [Background] Dorsch JA, Dorsch SE. Airway Equipment. In: Dorsch JA, Dorsch SE, editors. Understanding Anesthesia Equipment. 5th ed: Lippincott Williams and Wilkins; 2012. p. 593-8.
- [Background] Rosenbalt WH, Sukhupragarn W. Airway Management. In: Barash PG, Cullen BF, Stoeltin RK, Cahalan MK, Stock MC, Ortega R, editors. Clinical Anesthesia. 7th ed. Philadelphia: Lipincott Williams and Wilkins; 2013. p. 774-8.
- [Background] Connor CW. Commonly Used Monitoring Techniques. In: Barash PG, Cullen BF, Stoeltin RK, Cahalan MK, Stock MC, Ortega R, editors. Clinical Anesthesia. 7th ed. Philadelphia: Lippincott Williams and Wilkins; 2013. p. 704-6.
- [Background] Chitilian HV, Kaczka DW, Melo MFV. Respiratory Monitoring. In: Miller RD, Cohen NH, Eriksson LI, Fleisher LA, Wiener-Kronish JP, Young WL, editors. Miller's Anesthesia. 8th ed. Philadelphia: Elsevier Saunders; 2015. p. 1551-5.
- [Result] Chou HC, Tseng WP, Wang CH, Ma MH, Wang HP, Huang PC, Sim SS, Liao YC, Chen SY, Hsu CY, Yen ZS, Chang WT, Huang CH, Lien WC, Chen SC. Tracheal rapid ultrasound exam (T.R.U.E.) for confirming endotracheal tube placement during emergency intubation. Resuscitation. 2011 Oct;82(10):1279-84. doi: 10.1016/j.resuscitation.2011.05.016. Epub 2011 Jun 1. PMID 21684668
- [Result] Karacabey S, Sanri E, Gencer EG, Guneysel O. Tracheal ultrasonography and ultrasonographic lung sliding for confirming endotracheal tube placement: Speed and Reliability. Am J Emerg Med. 2016 Jun;34(6):953-6. doi: 10.1016/j.ajem.2016.01.027. Epub 2016 Jan 26. PMID 26994679
- [Result] Pfeiffer P, Rudolph SS, Borglum J, Isbye DL. Temporal comparison of ultrasound vs. auscultation and capnography in verification of endotracheal tube placement. Acta Anaesthesiol Scand. 2011 Nov;55(10):1190-5. doi: 10.1111/j.1399-6576.2011.02501.x. Epub 2011 Sep 8. PMID 22092123
- [Result] Das SK, Choupoo NS, Haldar R, Lahkar A. Transtracheal ultrasound for verification of endotracheal tube placement: a systematic review and meta-analysis. Can J Anaesth. 2015 Apr;62(4):413-23. doi: 10.1007/s12630-014-0301-z. Epub 2014 Dec 24. PMID 25537734
- [Result] Chou EH, Dickman E, Tsou PY, Tessaro M, Tsai YM, Ma MH, Lee CC, Marshall J. Ultrasonography for confirmation of endotracheal tube placement: a systematic review and meta-analysis. Resuscitation. 2015 May;90:97-103. doi: 10.1016/j.resuscitation.2015.02.013. Epub 2015 Feb 21. PMID 25711517
- [Result] Milling TJ, Jones M, Khan T, Tad-y D, Melniker LA, Bove J, Yarmush J, SchianodiCola J. Transtracheal 2-d ultrasound for identification of esophageal intubation. J Emerg Med. 2007 May;32(4):409-14. doi: 10.1016/j.jemermed.2006.08.022. Epub 2007 Apr 16. PMID 17499696
- [Result] Brun PM, Bessereau J, Cazes N, Querellou E, Chenaitia H. Lung ultrasound associated to capnography to verify correct endotracheal tube positioning in prehospital. Am J Emerg Med. 2012 Nov;30(9):2080.e5-6. doi: 10.1016/j.ajem.2011.10.023. Epub 2011 Dec 26. PMID 22205008
- [Result] Adi O, Chuan TW, Rishya M. A feasibility study on bedside upper airway ultrasonography compared to waveform capnography for verifying endotracheal tube location after intubation. Crit Ultrasound J. 2013 Jul 4;5(1):7. doi: 10.1186/2036-7902-5-7. PMID 23826756
- [Result] Li J. Capnography alone is imperfect for endotracheal tube placement confirmation during emergency intubation. J Emerg Med. 2001 Apr;20(3):223-9. doi: 10.1016/s0736-4679(00)00318-8. PMID 11267809
- [Result] Knapp S, Kofler J, Stoiser B, Thalhammer F, Burgmann H, Posch M, Hofbauer R, Stanzel M, Frass M. The assessment of four different methods to verify tracheal tube placement in the critical care setting. Anesth Analg. 1999 Apr;88(4):766-70. doi: 10.1097/00000539-199904000-00016. PMID 10195521
- [Result] Grmec S. Comparison of three different methods to confirm tracheal tube placement in emergency intubation. Intensive Care Med. 2002 Jun;28(6):701-4. doi: 10.1007/s00134-002-1290-x. Epub 2002 Apr 30. PMID 12107674
- [Result] Gottlieb M, Bailitz JM, Christian E, Russell FM, Ehrman RR, Khishfe B, Kogan A, Ross C. Accuracy of a novel ultrasound technique for confirmation of endotracheal intubation by expert and novice emergency physicians. West J Emerg Med. 2014 Nov;15(7):834-9. doi: 10.5811/westjem.22550.9.22550. Epub 2014 Nov 24. PMID 25493129
- [Result] Chou HC, Chong KM, Sim SS, Ma MH, Liu SH, Chen NC, Wu MC, Fu CM, Wang CH, Lee CC, Lien WC, Chen SC. Real-time tracheal ultrasonography for confirmation of endotracheal tube placement during cardiopulmonary resuscitation. Resuscitation. 2013 Dec;84(12):1708-12. doi: 10.1016/j.resuscitation.2013.06.018. Epub 2013 Jul 9. PMID 23851048
- [Result] Abhishek C, Munta K, Rao SM, Chandrasekhar CN. End-tidal capnography and upper airway ultrasonography in the rapid confirmation of endotracheal tube placement in patients requiring intubation for general anaesthesia. Indian J Anaesth. 2017 Jun;61(6):486-489. doi: 10.4103/ija.IJA_544_16. PMID 28655954

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT04316988/Prot_SAP_ICF_000.pdf